CLINICAL TRIAL: NCT01190670
Title: A Phase 1, Open Label, Drug Interaction Study of the Pharmacokinetics of ASP015K and Tacrolimus After Separate and Concomitant Administration to Healthy Adult Subjects
Brief Title: A Study to Evaluate the Drug Interaction of ASP015K and Tacrolimus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sr Manager Clinical Trials Registry, Astellas Pharma Global Development
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 015K-CL-PK16
Record Dates: First submitted 2010-08-11; First posted 2010-08-30 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Healthy; Pharmacokinetics of ASP015K and Tacrolimus
Keywords: ASP015K; tacrolimus; healthy volunteers
MeSH Terms: interventions — Tacrolimus; peficitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1, Group 1 (Experimental): ASP015K, low dose followed by high dose, with oral tacrolimus
  Interventions: Drug: Tacrolimus; Drug: ASP015K
- Part 1, Group 2 (Experimental): ASP015K, high dose followed by low dose, with oral tacrolimus
  Interventions: Drug: Tacrolimus; Drug: ASP015K
- Part 2 (Experimental): ASP015K high dose with intravenous tacrolimus
  Interventions: Drug: Tacrolimus; Drug: ASP015K

INTERVENTIONS:
Drug: Tacrolimus — Oral and Intravenous
  Other Names: FK506; Prograf
Drug: ASP015K — Oral

SUMMARY:
The objective of the study is to characterize the effect of multiple doses of ASP015K on the pharmacokinetics of a single oral dose or a single intravenous (IV) dose of tacrolimus.

DETAILED DESCRIPTION:
This is a 2-part study. Part 1 is a 2-sequence, drug interaction study to determine the effect of two different ASP015K doses on the pharmacokinetics of oral tacrolimus. Part 2 is a 1-sequence drug interaction study to determine the effect of the higher dose ASP015K on the pharmacokinetics of IV tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

* Subject weighing at least 45kg and body mass index (BMI) of 18-32 kg/m2, inclusive
* If female, subject is at least 2 years post menopausal or is surgically sterile per documentation provided by a third party medical professional and the subject is not pregnant as documented by a negative serum pregnancy test
* If male, subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy during the study period
* 12-lead ECG is normal or if abnormal, the abnormality is not clinically significant
* Clinical laboratory test results are within normal limits or not clinically significant
* Medically healthy, with no clinically significant medical history or abnormalities

Exclusion Criteria:

* History of any clinically significant disorder, disease or malignancy excluding non-melanoma skin cancer
* Recent history (within 6 months) of drug or alcohol abuse or positive urine screen for drugs of abuse/illegal drugs
* Treatment with prescription drugs or complementary and alternative medicines (CAM) within 14 days prior to study drug administration, or over the counter medication within 1 week prior to study drug administration
* A symptomatic, viral, bacterial or fungal infection within 1 week prior to clinic check-in
* Positive test for hepatitis C antibody, or positive test for hepatitis B surface antigen (HBsAg)
* History of human immunodeficiency virus (HIV) antibody
* Positive tuberculosis (TB) skin test or Quantiferon Gold test
* Vaccinated within the last 30 days prior to study drug administration
* Received an experimental agent within 30 days or five half-lives, whichever is longer, prior to study drug administration
* Any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission
* Absolute neutrophil count (ANC) <2500 cells/mm3

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables assessment through analysis of blood and urine samples | Days 1-13 and Days 26-33 (Part 1 only) sampled daily

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (1):
- Honolulu, Hawaii, United States